CLINICAL TRIAL: NCT03289754
Title: A Prospective Study to Evaluate the ConforMIS iTotal® (CR) Knee Replacement System and iPoly XE Tibial Inserts
Brief Title: A Prospective Study to Evaluate the iTotal Knee and iPoly XE Tibial Inserts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-001
Record Dates: First submitted 2017-09-15; First posted 2017-09-21 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee implant; osteoarthritis; patient-specific; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ConforMIS iTotal Knee with iPoly Insert (Experimental): The tibial insert being utilized in this study will be a highly-crosslinked, Vitamin-E enriched UHMWPE (iPoly XE) instead of traditional tibial inserts.
  Interventions: Device: iPoly XE tibial insert with ConforMIS iTotal KRS

INTERVENTIONS:
Device: iPoly XE tibial insert with ConforMIS iTotal KRS — The implants are constructed to conform to the surface of the patient's femoral condyle and proximal tibia, replacing the damaged cartilage with a smooth articulating surface. The femoral component and tibial tray are manufactured from cobalt chromium molybdenum alloy. The tibial insert and patellar component are manufactured from ultra-high molecular weight polyethylene.

SUMMARY:
This study is designed to evaluate the clinical outcomes of subjects who have recently undergone surgery with the iTotal® Cruciate Retaining (CR) Total Knee Replacement System (KRS) who have also had iPoly XE Tibial Inserts implanted.

DETAILED DESCRIPTION:
The study is prospective and single-center. Subjects will be implanted with an iTotal® CR Knee Replacement System in conjunction with an iPoly XE insert. The study will include a minimum of 50 subjects and a maximum of 60 subjects at a single center. The study site will be located in Germany. The study subjects will be followed for 10 years post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical condition included in the approved Indications For Use for the iTotal® CR
2. Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a TKR procedure. Disease status is assessed by Clinical and Radiographic assessment.
3. Willingness to participate in the clinical study, to give informed consent, and to attend all follow-up visits
4. > 18 years of age

Exclusion Criteria:

1. Simultaneous bilateral procedure required
2. BMI > 40
3. Active malignancy (defined as a history of any invasive malignancy - except non-melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
4. Poorly controlled diabetes
5. Neuromuscular conditions which prevent patient from participating in study activities
6. Active local or systemic infection
7. Immunocompromised
8. Fibromyalgia or other general body pain related condition
9. Rheumatoid arthritis or other forms of inflammatory joint disease
10. Loss of bone or musculature, osteonecrosis, neuromuscular or vascular compromise in the area of the joint to be operated on, to an extent that the procedure is unjustified
11. Diagnosed with or receiving treatment for Osteoporosis
12. Other physical disability affecting the hips, spine, or contralateral knee
13. Severe instability due to advanced loss of osteochondral structure
14. Prior arthroplasty of the affected knee, including High Tibial Osteotomy (HTO)
15. Compromised PCL or collateral ligament
16. Severe fixed valgus or varus deformity of >15º
17. Extensor lag > 15º
18. Fixed flexion contracture ≥ 15º
19. Unwilling or unable to comply with study requirements
20. Participation in another clinical study which would confound results
21. Allergy to any of the implant materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Drees, Principal Investigator — University- Mainz
Locations (1):
- University Medical Center of Johannes Gutenberg-University Mainz, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ConforMIS iTotal Knee With iPoly Insert
Started | 52
Completed | 49 (Study Terminated Early.)
Not Completed | 3
Not completed — Screen Failure or Failure to Meet Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Study terminated early.
Arm/Group | ConforMIS iTotal Knee With iPoly Insert
Number analyzed (Participants) | 49
Age, Continuous [Mean (Full Range); unit: years] — Population: The age of one patient who met screening criteria and follow-up duration did not have age reported.
  years
    number analyzed (Participants) | 48
    (all) | 66.27 [45 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient who met screening criteria and follow-up duration did not report sex.
  Participants
    number analyzed (Participants) | 48
    Female | 30
    Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 49

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Device-related Complications
Description: Adverse events were categorized as "Device Probably Related", "Device Possibly Related", Device All Related", or "Device Not Related" by the care team for all adverse events (as per the definitions of adverse events on clinicaltrials.gov). Outcome metrics are given in the form of "Events per Patient" which was calculated by dividing the number of adverse in each category by the number of baseline patients.
Time Frame: 1 year
Measure: Number; unit: Events per Patient
Groups:
- "Device Probably Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Device Probably Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Device Possibly Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Device Possibly Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Device All Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Device All Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Device Not Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Device Not Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
Arm/Group | "Device Probably Related" Adverse Event | "Device Possibly Related" Adverse Event | "Device All Related" Adverse Event | "Device Not Related" Adverse Event
Number analyzed (Participants) | 49 | 49 | 49 | 49
Events per Patient | 0.02 | 0.31 | 0.33 | 0.39

2. Primary Outcome: Incidence of Procedure-Related Complications
Description: Adverse events were categorized as "Procedure Probably Related", "Procedure Possibly Related", Procedure All Related", or "Procedure Not Related" by the care team for all adverse events (as per the definitions of adverse events on clinicaltrials.gov). Outcome metrics are given in the form of "Events per Patient" which was calculated by dividing the number of adverse in each category by the number of baseline patients.
Time Frame: 1 year
Measure: Number; unit: Events per Patient
Groups:
- "Procedure Probably Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Procedure Probably Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Procedure Possibly Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Procedure Possibly Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Procedure All Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Procedure All Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
- "Procedure Not Related" Adverse Event: Category of adverse event assigned by the care team indicating the likelihood of specific adverse events being considered "Procedure Not Related". Then, converted to "Event per Patient" to allow for simple comparison across different categories.
Arm/Group | "Procedure Probably Related" Adverse Event | "Procedure Possibly Related" Adverse Event | "Procedure All Related" Adverse Event | "Procedure Not Related" Adverse Event
Number analyzed (Participants) | 49 | 49 | 49 | 49
Events per Patient | 0.1 | 0.14 | 0.24 | 0.47

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from surgery date until 1 year post-operation.
Description: N/A. All reporting followed the definitions on clinicaltrials.gov
Arm/Group | ConforMIS iTotal Knee With iPoly Insert
All-Cause Mortality (participants affected / at risk) | 1/49
Serious Adverse Events (participants affected / at risk) | 15/49
Other Adverse Events (participants affected / at risk) | 12/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ConforMIS iTotal Knee With iPoly Insert (N=49)
Death (Congenital, familial and genetic disorders) | 1 (1) — Serious Adverse Event listed as "SAE_DEATH" by investigators
Life-threatening (General disorders) | 2 (2) — Events that posed an immediate risk to the patient's life requiring urgent intervention
Disability (General disorders) | 0 (0) — Events that resulted in persistent or significant disability or incapacity
Medical Intervention (General disorders) | 5 (7) — Events that required medical or surgical intervention to prevent death, life-threatening situations, or permanent disability.
Hospitalization (General disorders) | 7 (9) — Events that required inpatient hospitalization or prolonged existing hospitalization but did not meet other severity criteria
Other (General disorders) | 1 (1) — Serious adverse events that did not fit into standard severity categories or had incomplete severity documentation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ConforMIS iTotal Knee With iPoly Insert (N=49)
Infection Complications (Infections and infestations) | 3 (3)
Wound Infection (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombotic Complications (Vascular disorders) | 1 (1)
Pain/Stiffness Complications (General disorders) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT03289754/Prot_SAP_000.pdf